# **Cover letter**

| IN |
|--------------|
| ΙF |
| $\mathbf{O}$ |
| R |
| 1 |
| Æ |
| E |
| $\Gamma$ |
| ) |
| C |
| ( |
| )] |
| N |
| S |
| SI |
| 7 |
| N |
| Т |
| ٠. |
| F |
| )] |
| R |
| I |
| ) |
| 4 |
| R |
| ) [ |
| Γ |
| I( |
| 7 |
| H |
| ) |
| A |
| П |
| ` |
| ( |
| 1( |
| V |
| 1 |
| J |
| Δ |
| R |
| F |
| 3.5 |
| SI |
| Ξ. |
| A |
| F |
| 8 |
| C |
| F |
| Ŧ |
| S |
| Т |
| ľ |
| Л |
| D |
| 7 |
| 7 |

# **Official Study Title:**

Insertion of a Transoesophageal Echocardiography Probe Using the McGRATH Video Laryngoscope in Cardiac Surgery Patients: A Randomized Controlled Trial

ClinicalTrials.gov Identifier:

NCT number not yet assigned

**Document Type:** 

**Informed Consent Form** 

**Consent Form Version Date:** 

**January 7, 2026** 

#### INFORMED CONSENT FOR PARTICIPATION IN A RESEARCH STUDY

### **Study Title:**

Insertion of a Transoesophageal Echocardiography Probe Using McGRATH Video Laryngoscope in Cardiac Surgery Patients: A Prospective Randomized Study

### **Principal Investigator:**

Dr. Hassan Mohamed Ali

Professor of Anesthesia

Cairo University

#### Introduction

You are invited to participate in a research study. Before you decide whether to take part. It is important to understand the purpose of the study and what your participation will involve. Participation is voluntary and will not affect your medical care.

## **Purpose of the Study**

Insertion of a transoesophageal echocardiography (TEE) probe during cardiac surgery may cause injury to the pharynx or esophagus. The McGRATH video laryngoscope allows better visualization and may reduce these risks compared to the conventional technique.

## **Study Procedure**

The TEE probe will be inserted using a video laryngoscope during the scheduled surgical procedure only.

#### Risks

There is a very small risk of pharyngeal injury or temporary difficulty swallowing.

# Compensation

There are no financial compensation and no additional costs for participation.

### **Confidentiality**

All personal and medical information will be kept strictly confidential.

### **Voluntary Participation**

Participation is voluntary. You may withdraw at any time without affecting your care or legal rights.

# **Legal Rights**

Signing this informed consent form does **not** waive or limit any of your legal rights. It also does not release the researchers or the participating institution from their professional or legal responsibilities.

#### **Statement of Consent**

I have read and understood the information provided above. I have had the opportunity to ask questions, and all my questions have been answered satisfactorily. I voluntarily agree to participate in this research study.

| Participant Name (Print): | |
|---------------------------|-------|
| Participant Signature: | Date: |
| Researcher Signature: | Date: |